CLINICAL TRIAL: NCT00654550
Title: A Phase 1 Randomized, Prospective, Double-Masked, Vehicle-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability and Clinical Effect of Nexagon™ in Subjects Following Bilateral Photorefractive Keratectomy (PRK) for the Correction of Mild to Moderate Myopia.
Brief Title: A Study to Assess the Safety, Tolerability and Effect of Nexagon™ Applied to the Eye After PRK Laser Eye Surgery for Nearsightedness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OcuNexus Therapeutics, Inc. (Industry)
Responsible Party: Scott Bannan, CoDaTherapeutics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEX-OCU-001
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Corneal re-Epithelialization
Keywords: Photorefractive keratectomy; Re-epithelialization; Nexagon; PRK; Coda
MeSH Terms: conditions — Cavitary Optic Disc Anomalies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Nexagon™ or Nexagon™ vehicle

INTERVENTIONS:
Drug: Nexagon™ or Nexagon™ vehicle — Dose-escalation design in which cohorts of 6 subjects will be studied sequentially.

SUMMARY:
Phase 1 randomized, prospective, double-masked, vehicle-controlled, dose-escalation study to evaluate the safety, tolerability and clinical effect of Nexagon™ in subjects following bilateral PRK for the correction of mild to moderate myopia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pre-presbyopic myopes.
* Aged between 20 and 50 years inclusive.
* Females are eligible to participate only if they are currently non-pregnant and non-lactating. Females of child-bearing potential must commit to consistent and correct use of an acceptable method of birth control.
* Subjects willing and able to undergo bilateral PRK for the correction of their myopia.
* Subjects with MRSE <6.0 D, with less than 2.0 D of astigmatism.
* No more than 1.0 D of refractive difference between eyes.
* Stable prescription in both eyes as defined by <0.25 D change over the preceding 2 years.
* Subjects who are able to comply with all study procedures, including wearing a soft bandage contact lens in the immediate postoperative period.
* Subjects who are willing and able to give written informed consent to take part in the study.

Exclusion Criteria:

* Subjects who have a past or present disease, which as judged by the investigator may affect the safety of the subject or the outcome of the study.
* Subjects who have previously had corneal surgery.
* Subjects who require Mitomycin C following their PRK.
* Subjects with any ocular disease or corneal abnormality, including but not limited to:

  * Decreased corneal sensation / neurotrophic cornea;
  * Corneal vascularization;
  * Keratoconus;
  * Keratoconjunctivitis sicca requiring chronic treatment;
  * Lagophthalmos;
  * Blepharitis;
  * History of infectious keratitis;
  * History of glaucoma or intraocular pressure of >21 mmHg or use of glaucoma medications;
  * Significant dry eye disease that requires regular topical treatment;
  * Corneal thickness <480 µm at the thinnest point, and
  * Posterior elevation >40 mmHg.
* Subjects with corneal haze >+1 as assessed using the grading scale in the protocol.
* Subjects who require any topical ophthalmic medication other than the pre- and postoperative regimen defined in the study protocol.
* Subjects with:

  * Diabetes;
  * Collagen disorders associated with autoimmune diseases, e.g., lupus, rheumatoid arthritis;
  * Severe atopic disease;
  * Any systemic disease or condition where the subject is immunocompromized.
* Subjects who require any systemic medication that affects healing, e.g., steroids, hormone replacement therapy.
* Subjects who are taking amiodarone, long acting anticholinergics, e.g., atropine, scopolamine, or medications or agents that can cause dry eye.
* Subjects who have participated in a clinical trial within the 30 days prior to the date on which PRK is scheduled.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 30 days post-application

SECONDARY OUTCOMES:
To evaluate the clinical effect of Nexagon™ | 30 days post-application

CONTACTS AND LOCATIONS:
Overall Officials: Sue Ormonde, MD, FRC Ophth, FRANZCO, Principal Investigator — Auckland Eye
Locations (1):
- Auckland Eye Limited, Auckland, New Zealand